CLINICAL TRIAL: NCT03350295
Title: Open Label, Randomized, Single-dose, Cross-over Study to Evaluate the Relative Bioavailability, Safety, and Tolerability of Single Doses of Nifurtimox 30 mg Tablets Exhibiting Different in Vitro Dissolution Characteristics, and to Evaluate the Relative Bioavailability of Nifurtimox 30 mg and 120 mg Tablets, Administered to Adult Male and Female Patients With Chagas' Disease
Brief Title: Study Will Evaluate the Relative Bioavailability, Safety, and Tolerability of Single Doses of Nifurtimox 30 mg Tablets Exhibiting Different in Vitro Dissolution Characteristics, and to Evaluate the Relative Bioavailability of Nifurtimox 30 mg and 120 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16007
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Chagas Disease
Keywords: Relative bioavailability; In vitro dissolution
MeSH Terms: conditions — Chagas Disease | interventions — Nifurtimox

STUDY DESIGN:
Intervention Model Description: Group 1 ( Treatment A,B,C - 3 way cross-over), Group 2 ( Treatment D, E - 2 way cross over)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRP1 - Assess relative bioavailability(3-way cross-over) (Experimental): GROUP 1 (Treatments A, B, C) All 3 treatments in Group 1 consist of a dose of 120 mg nifurtimox (4 x 30 mg tablets). Participants received the 3 treatments in one of six treatment sequences under fed condition.
  Treatment A, dose administration with fast in vitro dissolution characteristics Treatment B, dose administration with medium in vitro dissolution characteristics Treatment C, dose administration with slow in vitro dissolution characteristics
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)
- GRP2 - Assess relative bioavailability (2-way cross-over) (Experimental): GROUP 2 (Treatments D and E) Participants received the 2 treatments in one of two treatment sequences under fed condition.
  Treatment D, a single dose 30 mg nifurtimox dose with medium in vitro dissolution characteristics Treatment E, a single dose of 120 mg nifurtimox
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)

INTERVENTIONS:
Drug: Nifurtimox (Lampit, BAYA2502) — Oral Intake of 4 x 30 mg nifurtimox tablets for treatment A-C; Oral Intake of 1 x 30 mg nifurtimox tablets for treatment D Oral intake of 1 x 120 mg nifurtimox tablet for treatment E

SUMMARY:
Study to assess the relative Bioavailability To assess the relative bioavailability of three formulations of nifurtimox 30 mg tablets exhibiting different in vitro dissolution profiles To assess the pharmacokinetics (PK) of nifurtimox To investigate the safety and tolerability of nifurtimox.

DETAILED DESCRIPTION:
Primary objective is to assess the relative bioavailability of three formulations of nifurtimox 30 mg tablets exhibiting different in vitro dissolution profiles (slow, medium, and fast, whereby "medium" represents the drug product currently used in clinical Phase 3 studies) under fed conditions in adult male and female patients with Chagas' disease.

A secondary objective of the study is to assess the relative bioavailability of nifurtimox after a single oral dose of 30 mg and 120 mg To assess the pharmacokinetics (PK) of nifurtimox To investigate the safety and tolerability of nifurtimox..

ELIGIBILITY:
Inclusion Criteria

* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and 12 weeks after the last administration of study drug. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements. Acceptable methods of contraception include, but are not limited to: (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception. Subjects must agree to utilize two reliable and acceptable methods of contraception simultaneously.
* Women of childbearing potential with confirmed last menstrual period by anamnesis and negative serum pregnancy test (beta-human chorionic gonadotropin [βhCG]) at screening and negative urine pregnancy test (βhCG) at pre-dose of each treatment.
* Women of non-childbearing potential, such as surgically sterile women with either written documentation of surgical sterility or negative serum pregnancy test (βhCG) at screening and negative urine pregnancy test (βhCG) at pre-dose of each treatment.
* Male subjects who agree not to act as sperm donors for 12 weeks after last administration of study drug.
* Age: 18 to 45 years (inclusive) at screening.
* Body mass index (BMI): ≥18 and <29.9 kg/m².
* Written informed consent must be provided before any study-specific tests or procedures are performed.
* Male/female patient diagnosed with chronic Chagas' disease:
* Previous diagnosis of acute or chronic Chagas' disease by a health clinic prior to screening for the study. The diagnosis of chronic Chagas' disease may be made by clinical findings, supported by antibody titers if available. If there is a known history of acute disease, it is preferable to have documentation of parasites on the blood smear, if available.

Exclusion Criteria

* Incompletely cured pre-existing diseases (except chronic Chagas' disease without active GI condition) for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study drugs will not be normal.
* Acute Chagas' disease. (During the acute phase, the parasite on a blood smear may be seen under a microscope. Different antibodies are present, depending on the course of the disease).
* Known hypersensitivity to the study drug (active substance or excipients of the preparations)
* Unstable or uncontrolled medical condition such as hypertension or diabetes, decompensated heart failure, GI conditions that would interfere with the absorption of the study drug (e.g. GI ulceration, peptic ulceration, GI bleeding, gastroesophageal reflux, or other GI disease affecting gastroesophageal junction), conditions that could potentially have an impact on drug metabolism or elimination (renal, hepatic such as known hepatic or biliary abnormalities), or any clinically relevant active infections in the opinion of the investigator within 4 weeks before the screening visit, e.g. clinically relevant history or presence of significant respiratory (e.g. interstitial lung disease), hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic (e.g. diabetes), and dermatological or connective tissue disease.
* Use of systemic or topical medicines or substances which oppose the study objectives (including clinical treatment with nifurtimox and benznidazole) or which might influence them within 4 weeks before the first study drug administration, e.g. an investigational drug, any drug altering GI motility and/or gastric pH (e.g. antacids, anticholinergic, para-sympatholytics), any drug known to induce liver enzymes (e.g. dexamethasone, barbiturates, St. John's Wort [hypericum perforatum]), any drug known to inhibit liver enzymes (e.g. ketoconazole, macrolides).
* Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over 120 msec or of the QT interval over 450 msec using Bazett's formula (QTcB). (Clinically stable subjects with Chagas'-related heart disease and pacemaker in place for >1 year and evaluated by a cardiologist ≤6 months before the first dose of study drug will not be excluded.)
* Systolic blood pressure <100 or >140 mmHg (after resting in supine position for a minimum of 3 minutes).
* Diastolic blood pressure <50 or >90 mmHg (after resting in supine position for a minimum of 3 minutes).
* Findings that would exclude the subject in the investigator's judgment, e.g. enlarged liver, irregular heartbeat, undiagnosed acute illness, and melanoma.
* Positive pregnancy test.
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV 1+2).
* Positive urine drug screening..

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlast) of nifurtimox | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  AUC(0-tlast):Area under the drug-concentration vs. time curve of nifurtimox from time 0 to the last data point
Cmax of nifurtimox | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration
AUC of nifurtimox | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
  AUC: Area under the concentration versus time curve from zero to infinity after single (first) dose

SECONDARY OUTCOMES:
Number of participants with adverse events | up to 8 weeks
AUC divided by dose: AUC/D | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
AUC(0-tlast) divided by dose: AUC(0-tlast)/D | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour
Cmax divided by dose: Cmax/D | 0, 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12,15 hour

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- FP Clinical Pharma, Buenos Aires, Ciudad Auton. de Buenos Aires, Argentina

REFERENCES:
- [Derived] Stass H, Just S, Weimann B, Ince I, Willmann S, Feleder E, Freitas C, Yerino G, Munster U. Clinical investigation of the biopharmaceutical characteristics of nifurtimox tablets - Implications for quality control and application. Eur J Pharm Sci. 2021 Nov 1;166:105940. doi: 10.1016/j.ejps.2021.105940. Epub 2021 Jul 12. PMID 34265407